CLINICAL TRIAL: NCT04135287
Title: Relationship Between Improvement in Insulin Secretion and Decrease in HbA1c in GLP-1 RA Therapy in T2DM Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA HM-2019-004
Record Dates: First submitted 2019-10-20; First posted 2019-10-22 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: GLP-1 RA
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to receive for 6 months in an open label fashion GLP1RA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Treatment with GLP-1 RA
  Interventions: Drug: GLP-1 receptor agonist

INTERVENTIONS:
Drug: GLP-1 receptor agonist — The main objective of the study is to determine the relationship between the increase in glucose-stimulated insulin secretion and decrease in HbA1c caused by GLP-1 RA therapy in poorly controlled T2DM patients. We also will identify a cut point of an increase in beta cell function which produces a clinically meaningful decrease in HbA1c.

SUMMARY:
GLP-1 receptor agonists (GLP-1 RA) is group of antidiabetic agents very effective in lowering the plasma glucose concentration in T2DM patients . Currently there are several agents approved for the treatment of T2DM which are classified into two groups: (1) short acting GLP-1 RA and include exenatide BID and lexisenatide, and (2) long acting agents which are given once daily or weekly injection and include liraglutide, semaglutide, dulaglutide and budyreon . Clinical studies have demonstrated that long acting GLP-1 RA (e.g. liraglutide, bydureon and dulaglutide) produce ~1.5% reduction in the HbA1c , which was significantly greater than that caused by other classes of antidiabetic agents (e.g. DPP4 inhibitors, and SGLT2 inhibitors). Members of this class of drugs exert multiple metabolic actions in T2DM. They potentiate insulin-stimulated insulin secretion from the beta cell , inhibit glucagon secretion from the alpha cells and inhibit appetite and promote weight loss. Together, these metabolic actions of GLP-1 RA contribute to the improvement in glucose metabolism and decrease in HbA1c.

Although GLP-1 RA produce a robust mean decrease in HbA1c (~1.5%), the magnitude of decrease in HbA1c in the individual patient vary considerably. Clinical studies showed that approximately one third of T2DM patients receiving GLP-1 RA experience very modest to no decrease in the HbA1c while another third of patients experience a robust decrease in the HbA1c. the reason for this large variability in the individual response to GLP-1 RA is unknown. Studies which attempted to identify possible clinical predictors that distinguish between "good responders" and "poor responders" have failed to identify clinical parameter that can predict the magnitude of decrease in HbA1c by GLP-1 RA in T2DM patients.

Because of the central role of beta cell function in the regulation of plasma glucose concentration, the study investigators hypothesis that varying degree of beta cell response to GLP-1 RA action is the principal factor responsible for the large variability in the decrease in HbA1c by GLP-1 RA. The aim of the present study is to test this hypothesis.

DETAILED DESCRIPTION:
Study Design: Eligible subjects will receive the following: (1) medical history and physical examination, (2) Measurement of general chemistry, CBC, HbA1c, TSH, and (3) 75 grams OGTT.

After completing the OGTT, subjects will be randomized to receive for 6 months, in an open label fashion: (1) weekly exenatide (bydureon) 2 mg per week (n=105); (2) liraglutide 1.8 mg per day (n=105); or (3) dulaglutide 1.5 mg per week (n=105).

Liraglutide will be started on 0.6 mg/day and dulaglutide will be started at 0.75 mg/week and the dose will be increased to the maximal tolerated dose according to the patient response.

During the treatment period, subjects will be seen monthly for follow-up visits. Each visit, medical history, physical examination will be performed. Body weight, blood pressure, FPG, Insulin, C-Peptide, glucagon, and HbA1c will be measured. At the end of 6-month treatment period, the OGTT will be repeated.

Patient will be asked to bring the injection device at each monthly follow-up visit, and patient's compliance will be examined. Subjects with compliance rate <80% will be dropped off the study by the PI and other patient will be recruited to replace him

MATERIAL AND METHODS Screening: During this visit a complete medical history and physical exam will be performed. Blood will be drawn for general chemistries, lipid profile, complete blood count (CBC), and thyroid function tests (TSH and T3, T4). An additional 30 ml blood will be drawn and immediately frozen for the measurement of adipocytokines (adiponectin, TNF-alpha, IL6, resistin, leptin and hsCRP) and DNA extraction.

OGTT: All subjects will receive a 75 gram OGTT at 0800h after a 10-12 h overnight fast. Plasma glucose, insulin, C-peptide, GLP-1, GIP, glucagon, and FFA concentrations are measured at baseline (-15, -10 and 0 min) and every 30 min for 2 hours after glucose ingestion. Insulin sensitivity is calculated using the Matsuda Index (MI) of insulin sensitivity, which agrees closely with that measured with the euglycemic insulin clamp technique. The following indices of insulin secretion will be measured: early insulin response (ΔI0-30/ΔG0-30; ΔC-Pep0-30/ΔG0-30; ΔISR0-30/ΔG0-30) and total insulin response (ΔI0-120/ΔG0-120; ΔC-Pep0-120/ΔG0-120; ΔISR0-120/ΔG0-120), where ISR = insulin secretory rate calculated by plasma C-peptide deconvolution. Beta cell function is assessed using the insulin secretion/insulin resistance (disposition) index and is calculated as (ΔI/ΔG x Matsuda index; ΔISR/ΔG x Matsuda index).

Beta cell function during the OGTT also will be assessed using the Mari-Ferrannini model. This model expresses insulin secretion (in pmol min-1m-2) as the sum of two components: (i) beta cell glucose sensitivity which represents the dependence of insulin secretion on the plasma glucose concentration at any time point during the OGTT; (ii) rate sensitivity which represents the dependence of insulin secretion on the rate of change of plasma glucose. The ISR-plasma glucose dose-response curve is modulated by a potentiation factor that encompasses several potentiating mechanisms (prolonged exposure to hyperglycemia, non-glucose substrates, gastrointestinal hormones, neural modulation, time-dependent molecular/biochemical/enzymatic changes within the beta cell). In normal individuals, the potentiation factor typically increases from baseline to the end of the OGTT.

During the OGTT, 20 ml blood will be drawn to extract DNA and genome wide association analysis will be performed to identify genetic markers associated with beta cell function.

ELIGIBILITY:
Inclusion Criteria:

1. age 21-75 years
2. BMI=18-45 kg/m2
3. HbA1c >7.% and <14.0%
4. Subjects must be on stable antihyperglycemic therapy during the 3 months prior to enrolment.
5. Good general health as determined by physical exam, medical history, blood chemistries, CBC, TSH, T4, lipid profile.
6. Stable body weight (± 3 lbs) over the preceding three months
7. Not participate in an excessively heavy exercise program.

Exclusion Criteria:

1. Subjects receiving therapy with GLP-1 RA or received in the past 3 months. Subjects who received GLP-1 therapy > 3 months prior to the study are eligible to participate if their body weight has returned to the pretreatment level.
2. Subjects receiving DPP4 inhibitors or who received DPP4 inhibitor in the 3 month preceding the study. Subjects on DPP4 inhibitors who are interested in switching therapy to GLP-1 RA must have 3 months washout period.
3. Haematocrit < 32.0
4. history of thyroid cancer or pancreatitis,
5. Creatinine > 1.5 mg/dl,
6. history of malignant disease,
7. Pregnancy.
8. Congestive heart failure

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 6 months
  Change in HbA1c from baseline to 6 months

SECONDARY OUTCOMES:
Beta cell function | 6 months
  Change in Beta cell function measured as ∆C-Pep/(∆G/IR) and glucose sensitivity during OGTT
Weight loss | 6 months
  Change in body weight from baseline to 6 months
Fasting Plasma Glucagon | 6 months
  Change in FPG from baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa AlOzairi, MD, PhD, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait